CLINICAL TRIAL: NCT01487772
Title: Improving Quality of Care for Hip-Fracture Patients: Studies on Fast-track Surgery
Acronym: Q-HIP
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Consultant Orthopaedic Surgeon, Danderyd Hospital
Other Study IDs: 2010/685-32
Record Dates: First submitted 2011-12-06; First posted 2011-12-07 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip-fracture patients: Hip-fracture patients admitted to Orthopaedic Department of Danderyd Hospital

SUMMARY:
The aims of the studies are to examine the impact of delayed time to surgery for hip-fracture patients with regard to in-hospital complication rate and one-year mortality and to evaluate two different fast-track systems for hip-fracture patients with regard to patient outcome, complication rate and patient satisfaction.

DETAILED DESCRIPTION:
The aims of the studies are to examine the impact of delayed time to surgery for hip-fracture patients with regard to in-hospital complication rate and one-year mortality and to evaluate two different fast-track systems, the hip process pathway and the ambulance process pathway, for hip-fracture patients with regard to patient outcome, complication rate and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture

Exclusion Criteria:

* Periprosthetic fractures
* Pathological fractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hip-fracture patients admitted to the Orthopaedic Department of Danderyd Hospital during a two-year period.
Sampling Method: Non-Probability Sample
Enrollment: 1307 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Complication rate | 3-months
  The 3-month medical complication rate

SECONDARY OUTCOMES:
Mortality rate | 1-year
  One-year mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Olof Skoldenebrg, MD, PhD, Principal Investigator — Danderyd Hospital, Stockholm, Sweden
Locations (1):
- Danderyd Hospital, Stockholm, Sweden